CLINICAL TRIAL: NCT03041532
Title: Impact of Proximal Colon Retroflexion in Colorectal Cancer Screening Programme: Randomized Trial
Brief Title: Impact of Proximal Colon Retroflexion in Colorectal Cancer Screening Programme
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital del Rio Hortega (Other)
Responsible Party: Principal Investigator, Mª Henar Núñez Rodriguez, Principal Investigator: Dra Mª Henar Núñez Rodriguez, Hospital del Rio Hortega
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: CEIC 62/16
Record Dates: First submitted 2017-01-25; First posted 2017-02-02 (Estimated); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Colorectal Neoplasms; Adenoma Detection Rate
Keywords: retroflexion proximal; colorectal cancer screening programme; adenoma detection rate; right colon
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- proximal retroflexion (Experimental): Procedure: The endoscopy explore right colon with frontal view and a second look with proximal retroflexion
  Interventions: Procedure: Proximal retroflexion; Procedure: Frontal view
- frontal view of right colon (Active Comparator): Procedure: The endoscopy explore right colon with frontal view and frontal view
  Interventions: Procedure: Frontal view

INTERVENTIONS:
Procedure: Proximal retroflexion — The investigator explore twice right colon, first front view and second forward viewing or proximal retroflexion depends on randomization
  Arms: proximal retroflexion
Procedure: Frontal view — The investigator explore twice right colon with frontal viewing

SUMMARY:
Colorectal cancer (CRC) is the most common tumor and the second leading cause of death in the Western world. The decrease in incidence and mortality by CRC in the population undergoing screening has been observed. Colonoscopy is the recommended method for detecting tumors in early stages, as well as identifying and resecting adenomatous polyps, which are the precursor lesions of most CRCs. Colonoscopy should be of high quality to decrease incidence and mortality by CRC and avoid interval cancer. The literature shows that colonoscopy does not prevent right colon lesions in the same way as the left colon lesions, with most of the interval cancers located in the right colon. Studies published so far show an increase in the adenomas detection rate (ADT) in the right colon in the second visualization of this segment and an increase between 2 and 10% if this second examination is performed with the proximal retroflexion maneuver.Retroflexion is a safe maneuver in expert endoscopists. The aim of our study is to evaluate the ADT in the right colon by means of a second visualization by performing proximal retroflexion or second frontal visualization at random in the CCR screening population.

ELIGIBILITY:
Inclusion Criteria:

* Subjects participating in the Colorectal cancer Screening program with faecal immunological test > 100ng / ml.
* Ages between 50-69 years.
* Adequate preparation according to the Boston scale: in right colon (score> 2 in this section)
* Informed consent.

Exclusion Criteria:

* Refusal to give informed consent.
* Subjects with elevated colorectal cancer risk due to family history or inherited diseases of polyposis or inflammatory bowel disease
* Symptomatic subjects.
* Diverticulitis, inflammatory bowel disease or colonic stenosis during the exploration
* Inadequate preparation according to Boston cleanliness scale (score ≤ 2 in right colon)

Ages: 50 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 692 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Proximal retroflexion improve adenoma detection rate in colorectal cancer screening | through study completion, an average of 1 year
  Determine whether to perform retroflexion proximal improves adenoma detection rate in the right colon versus forward vision in population screening colorectal cancer with medium risk with immune blood test positive stool

SECONDARY OUTCOMES:
Second look for right colon improve adenoma detection rate | through study completion, an average of 1 year
  Determine if a second look: retroflexion proximal or forward view improve adenoma detection rate
Rate of retroflexion related adverse events | through study completion, an average of 1 year
Rate of retroflexion proximal adverse events with a pediatric colonoscopy | through study completion, an average of 1 year
Pre-procedure factors | through study completion, an average of 1 year
  To analyze pre-procedure factors that may influence the prevalence of precursor lesions in the colon: age, sex, race, alcohol, smoking habit and the value of SOH, in which more detailed explorations should be performed using proximal retroflexion

CONTACTS AND LOCATIONS:
Overall Officials: Mª Henar Núñez Rodriguez, Principal Investigator — Hospital del Rio Hortega Valladolid, Spain
Locations (1):
- Hospital Universitario Rio Hortega, Valladolid, Spain